CLINICAL TRIAL: NCT02396108
Title: Phase Ib Dose-confirmation Study of ASLAN001 Combined With Weekly Paclitaxel and Carboplatin in Advanced Solid Tumours, Followed by an Open-label Phase II Study in Patients With Stage I-III HER2 Positive Breast Cancer
Brief Title: Dose-confirmation Study of ASLAN001 Combined With Weekly Paclitaxel and Carboplatin in Advanced Solid Tumours, Followed by a Study in Patients With Stage I-III HER2 Positive Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014/01282
Record Dates: First submitted 2015-02-15; First posted 2015-03-24 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel + Carboplatin + ASLAN001 (Experimental): Phase I:
  A modified 3+3 study de-escalating dose design will be employed for dose determination. Subjects will receive treatment in 21-day cycles until disease progression, intolerable toxicities or withdraws consent. In the presence of intolerable toxicities to one or more of the drugs in the regimen (but not all 3), the drug in question may be discontinued and the other drugs continued with the patient remaining in the study, if the patient is deemed to be benefiting, after discussion with the Principal Investigator.
  Phase II:
  Patients with stage I-III HER2-positive breast cancer with a primary breast tumour of 2cm or greater will receive up to 4 cycles of pre-operative ASLAN001 and weekly paclitaxel/ carboplatin delivered in 21-day cycles. Prior to administration of chemotherapy, there will be lead-in dosing of single-agent ASLAN001 administered daily for 2 weeks at the recommended phase II dose.
  Interventions: Drug: Paclitaxel + Carboplatin + ASLAN001

INTERVENTIONS:
Drug: Paclitaxel + Carboplatin + ASLAN001 — Phase I
  * IV Paclitaxel 80mg/m2, day 1, 8, 15 of a 21-day cycle
  * IV Carboplatin AUC of 1.5, day 1, 8, 15 of a 21-day cycle
  * PO ASLAN001 daily continuously (starting dose 500mg BID)
  Phase II
  •PO ASLAN 001 daily continuously at the recommended phase II dose x 2 weeks
  Followed by:
  * IV Paclitaxel 80mg/m2, day 1, 8, 15 of a 21-day cycle x 4 cycles
  * IV Carboplatin AUC of 1.5, day 1, 8, 15 of a 21-day cycle x 4 cycles
  * PO ASLAN001 daily continuously at the recommended phase II dose x 12 weeks

SUMMARY:
The current standard of care for stage I-III HER2-positive breast cancer is adjuvant chemotherapy combined with 1 year of adjuvant trastuzumab. Neoadjuvant chemotherapy in early stage breast cancer has the advantages of i) tumour downsizing, ii) higher breast conservation rates, and iii) enabling the evaluation of tumour biology. Pathologic complete response following neoadjuvant chemotherapy has been shown to be an independent, strong predictor of outcome in operable HER2-positive breast cancer. The addition of neoadjuvant anti-HER2 therapy to chemotherapy results in a 2-3 fold increase in pCR rates in operable HER2-positive breast cancer. However, the optimal neoadjuvant regimen has not been defined in HER2-positive breast cancer. The investigators recently completed a phase II study of neoadjuvant lapatinib combined with weekly paclitaxel/ carboplatin in stage I-III HER2-positive breast cancer. Preliminary analysis suggested that the utility of the regimen might have been limited by its unfavourable efficacy/ toxicity ratio. ASLAN001 is a small molecule tyrosine kinase inhibitor against HER1, HER2, and HER4. Preclinical data have shown ASLAN001 to be more potent than lapatinib and neratinib in inhibiting HER1 and HER2, and early phase clinical studies have demonstrated superior pharmacokinetics and pharmacodynamic target inhibition compared to lapatinib. Furthermore, ASLAN001 has demonstrated a better safety profile than lapatinib in early phase studies.

• The investigators hypothesize that ASLAN001 combined with paclitaxel/carboplatin will induce favorable pathological complete response (of at least 30%) in stage I-III HER2 positive breast cancer, with a more favourable safety profile than lapatinib combined with paclitaxel/carboplatin.

DETAILED DESCRIPTION:
Breast cancer is the leading cause of cancer death among women worldwide, with approximately 800, 000 breast cancer deaths annually projected to occur in 2030 globally[1]. Activation and over-expression of oncogenes encoding trans-membrane receptor tyrosine kinases of the epidermal growth factor receptor (EGFR) family, including ErbB1 (also known as HER1/EGFR) and ErbB2 (also known as human epidermal growth factor receptor 2 or HER2), play an important role in the development of breast cancer. Overexpression of HER2 has been shown to be a poor prognostic indicator associated with increased relapse rates and poorer overall survival in breast cancer. Several therapeutic strategies have been developed to block HER2 signaling pathways in order to improve the treatment of breast cancer.

Trastuzumab is a recombinant, humanized, monoclonal antibody that binds to the extracellular domain of the HER2 protein. Treatment with trastuzumab improves the outcomes of women with HER2 over-expressing early stage and metastatic breast cancer (MBC) [3, 4]. The current standard of care for stage I-III HER2-positive breast cancer patients is the addition of 1 year of adjuvant trastuzumab to chemotherapy [5]. This results in a 40-50% improvement in 5- year disease-free survival (DFS), and 30% improvement in 5-year overall survival (OS) over chemotherapy alone.

Preoperative (primary or neoadjuvant) chemotherapy which is the standard therapy for patients with locally advanced breast cancer, is increasingly used in patients with operable breast cancer [15]. Randomised trials comparing preoperative and adjuvant chemotherapy for early operable breast cancer demonstrated that preoperative chemotherapy has several potential advantages over the adjuvant approach. It significantly increased the rate of breast conserving surgery over mastectomy. Pathological complete response following preoperative chemotherapy in the breast and lymph nodes significantly predicted better patient survival. Furthermore, preoperative chemotherapy was associated with fewer adverse events (AEs) [16, 17].

These data have prompted the increasing use of preoperative chemotherapy in patients with operable breast cancer. Given the increasingly important role of anti-HER2 therapy in both early and advanced stage HER2-positive breast cancer, our aim is to expand current therapeutic options by developing an efficacious and tolerable combination of chemotherapy and targeted therapy. In the neoadjuvant setting, the addition of trastuzumab to chemotherapy has been reported to result in a 2-3 fold increase in pCR rates in operable HER2-positive breast cancer [18].

However, the optimal neoadjuvant regimen for early stage HER2-positive breast cancer has yet to be defined. We recently completed a phase II study of neoadjuvant weekly paclitaxel and carboplatin in combination with lapatinib in patients with stage I-III HER2-positive breast cancer. Pathologic complete response rates were lower than expected (11.1%) due to a high proportion of locally advanced tumours. In addition, dose interruptions and reductions were common, and dose intensity was difficult to maintain. Grade 3 and above non-hematologic toxicities occurred in 19.4% and common toxicities (¬>20%) included diarrhea (80%), peripheral neuropathy (65.7%), rash (57.1%), nausea (40%), fatigue (40%), vomiting (34.3%), non-neutropenic infections (25%) and transaminitis (22.8%) [19]. ASLAN001 is a small molecule tyrosine kinase inhibitor against HER1, HER2, and HER4.

Preclinical data have shown ASLAN001 to be more potent than lapatinib and neratinib in inhibiting HER1 and HER2, and early phase clinical studies have demonstrated superior pharmacokinetics and pharmacodynamic target inhibition compared to lapatinib. Furthermore, ASLAN001 has demonstrated a better safety profile than lapatinib in early phase studies. We hypothesize that the novel combination of ASLAN001 with weekly paclitaxel/carboplatin will induce favorable pathological complete response (of at least 30%) in stage I-III HER2 positive breast cancer, with a more favourable safety profile than lapatinib combined with paclitaxel/carboplatin. All patients will receive 1 year of adjuvant trastuzumab following completion of anthracycline-containing chemotherapy post-operatively, in accordance with standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years
* Karnofsky performance status of 70 or higher
* Estimated life expectancy of at least 12 weeks
* Adequate organ function including the following:

Bone marrow:

oAbsolute neutrophil (segmented and bands) count (ANC) ≥ 1.5 x 109/L oPlatelets ≥ 100 x 109/L

Hepatic:

oBilirubin ≤ 1.5 x upper limit of normal (ULN), oALT and AST ≤ 2.5x ULN

Renal:

oCalculated creatinine clearance >30ml/minute

* Left ventricular ejection fraction ≥50% measured by 2D echo or MUGA
* Signed informed consent from patient or legal representative
* Patient with reproductive potential must use an approved contraceptive method if appropriate (e.g. intrauterine device, birth control pills, or barrier device) during and for three months after the study. Females with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment

Specific to phase I:

•Any patient with advanced cancer where treatment with weekly paclitaxel/ carboplatin is indicated, as determined by his/her physician

Specific to phase II:

* Histologic or cytologic diagnosis of breast carcinoma
* T1-4 breast cancer with measurable primary breast tumor, defined as palpable tumor with the largest diameter measuring 2.0cm or greater by calipers. For T1 breast cancer, the primary tumor must measure at least 2.0cm
* Tumor is HER2 positive either by IHC (3+) or FISH amplification (amplification ratio >2.0)

Exclusion Criteria:

* Concurrent administration of any other tumor therapy, including cytotoxic chemotherapy, endocrine therapy, and immunotherapy
* Major surgery within 28 days of study drug administration
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy
* Breast feeding
* Serious cardiac illness or medical conditions including but not confined to:

oHistory of documented congestive cardiac failure or systolic dysfunction (LVEF <50%) oHigh-risk uncontrolled arrhythmias (ventricular tachycardia, high-grade AV block, supraventricular arrhythmias which are not adequately rate-controlled) oHistory of significant ischaemic heart disease oClinically significant valvular heart disease oPoorly controlled hypertension (e.g. systolic BP > 180mmHg or diastolic >100mmHg)

* Poorly controlled diabetes mellitus.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* History of significant neurological or mental disorder, including seizures or dementia.
* Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones or stable chronic liver disease per investigator assessment)

Specific to phase I:

•Treatment with anti-tumour therapy, defined as chemotherapy, immunotherapy or investigational product within 21 days prior to first dose of study drug

Specific to phase II:

* Stage IV breast cancer
* Stage I breast cancer with primary breast tumor measuring <2.0cm
* Treatment within the last 28 days with any investigational drug

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response rate | Post neoadjuvant chemotherapy (within 2-3 weeks after last dose of neoadjuvant chemotherapy)
  Defined as the absence of invasive cancer in both the primary tumor as well as the axillary lymph nodes at the time of surgical resection.

SECONDARY OUTCOMES:
Treatment related toxicities, using descriptive statistics | Until death or disease progression, whichever occurs first (up to 5 years)
  Adverse events of special interest include febrile neutropenia, diarrhea, hepatotoxicity, and left ventricular dysfunction.
Breast conservation rates, using descriptive statistics | Post neoadjuvant chemotherapy (within 2-3 weeks after last dose of neoadjuvant chemotherapy)
  Odds ratio with approximate 95% confidence intervals for mastectomy (vs breast conservation) will be calculated for clinico-pathological factors known to influence breast surgery outcome following neoadjuvant chemotherapy, including clinical T and N stage at diagnosis, hormone receptor status, age (>40 vs ≤40) , and clinical response to chemotherapy.
Clinical response rate, using descriptive statistics | Post neoadjuvant chemotherapy (within 2-3 weeks after last dose of neoadjuvant chemotherapy)
  Will be calculated as the ratio of the number of complete and partial responders to the total number of evaluable patients, on completion of neoadjuvant chemotherapy. The response will be determined according to the RECIST criteria. A 80% confidential interval for the response rate will be computed based on the binomial distribution function. Waterfall plots will be constructed to visualize the extent of tumor regression after completing neoadjuvant chemotherapy and prior to surgery.
Relapse free survival (RFS), using Kaplan Meier/ log-rank test | 2 and 5 year post neoadjuvant chemotherapy/time of surgery
  Kaplan Meier curves of RFS at 2 and 5 years, of the entire cohort, the cohort that achieves pathological complete response and the cohort that does not achieve pathological complete response, will be plotted. Log-rank testing will be performed to identify clinical and pathological factors that influence RFS.
Identification of tumor biomarkers, using chi-square | Post neoadjuvant chemotherapy (within 2-3 weeks after last dose of neoadjuvant chemotherapy)
  Correlative testing of potential tumour biomarkers with presence or absence of pCR.

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Wong A, Tan SH, Soh T, Tan CS. Phase II study of neoadjuvant weekly paclitaxel and carboplatin with lapatinib in HER2+ breast cancer. J Clin Oncol 32:5s, (suppl; abstr 619), 2014.
- [Background] Romond EH, Perez EA, Bryant J, Suman VJ, Geyer CE Jr, Davidson NE, Tan-Chiu E, Martino S, Paik S, Kaufman PA, Swain SM, Pisansky TM, Fehrenbacher L, Kutteh LA, Vogel VG, Visscher DW, Yothers G, Jenkins RB, Brown AM, Dakhil SR, Mamounas EP, Lingle WL, Klein PM, Ingle JN, Wolmark N. Trastuzumab plus adjuvant chemotherapy for operable HER2-positive breast cancer. N Engl J Med. 2005 Oct 20;353(16):1673-84. doi: 10.1056/NEJMoa052122. PMID 16236738
- [Background] Perez EA, Romond EH, Suman VJ, Jeong JH, Davidson NE, Geyer CE Jr, Martino S, Mamounas EP, Kaufman PA, Wolmark N. Four-year follow-up of trastuzumab plus adjuvant chemotherapy for operable human epidermal growth factor receptor 2-positive breast cancer: joint analysis of data from NCCTG N9831 and NSABP B-31. J Clin Oncol. 2011 Sep 1;29(25):3366-73. doi: 10.1200/JCO.2011.35.0868. Epub 2011 Jul 18. PMID 21768458
- [Derived] Lee MX, Wong ALA, Ow S, Sundar R, Tan DSP, Soo RA, Chee CE, Lim JSJ, Yong WP, Lim SE, Goh BC, Wang L, Lee SC. Phase Ib Dose-Finding Study of Varlitinib Combined with Weekly Paclitaxel With or Without Carboplatin +/- Trastuzumab in Advanced Solid Tumors. Target Oncol. 2022 Mar;17(2):141-151. doi: 10.1007/s11523-022-00867-0. Epub 2022 Feb 23. PMID 35195837